CLINICAL TRIAL: NCT00938236
Title: CIS002: An Open-Label, Multi-Center, Extension Study of Cyclosporine Inhalation Solution in Subjects Previously Enrolled in the APT Study CIS001
Brief Title: CIS001 Extension Study of Cyclosporine Inhalation Solution
Acronym: CIS002
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Parent study CIS001 was completed
Sponsor: APT Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CIS002
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-09

CONDITIONS: Lung Transplant
Keywords: lung transplant; lung transplant recipient; bronchiolitis obliterans syndrome; bronchiolitis obliterans; single lung transplant; double lung transplant; heart-lung transplant; Aerosol
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Bronchiolitis Obliterans

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Inhaled cyclosporine (Other): Extended access to inhaled cyclosporine for patients from treatment and control arms of Phase 3 study CIS001
  Interventions: Drug: Cyclosporine Inhalation Solution (CIS)

INTERVENTIONS:
Drug: Cyclosporine Inhalation Solution (CIS) — Cyclosporine (USP) Inhalation Solution; 300mg/4.8 mL in propylene glycol (USP) at a concentration of 62.5 mg/mL; 3 times a week for study duration

SUMMARY:
This trial is a longterm follow up of a phase III study of inhaled cyclosporine for the prevention of chronic rejection in lung transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

1. Enrollment in study CIS001
2. Written informed consent for CIS002
3. Use of an effective means of contraception by women of childbearing potential

Exclusion Criteria:

1. Any unresolved or irreversible CIS-related ongoing serious adverse event
2. Subjects who have developed newly emergent conditions, injuries, diagnoses, physical examination findings, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk of treatment complications
3. Subjects with suspected or documented allergy to propylene glycol and/or cyclosporine
4. Women who are pregnant, wishing to become pregnant, or unwilling to use appropriate birth control to avoid becoming pregnant
5. Women who are breastfeeding
6. Subjects unable to comply with all protocol requirements and follow-up procedures
7. Subjects who discontinued from CIS002 to participate in another clinical trial and have received any investigational treatment (other than CIS) within 14 days of titration visit 1/baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-12; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To assess the long-term safety of CIS administration | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bruce A Johnson, MD, Principal Investigator — University of Pittsburgh; Jeffrey Golden, MD, Principal Investigator — University of California, San Francisco
Locations (16):
- United States (15):
  - UCLA School of Medicine, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado Health Sciences Cente, Denver, Colorado
  - University of Florida Health Sciences Center, Gainesville, Florida
  - Tampa General Hospital, Tampa, Florida
  - Loyola University Hospital, Maywood, Illinois
  - Indiana Methodist Research Institute, Indianapolis, Indiana
  - University of Maryland, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - New York Presbyterian Hospital, Columbia University Med. Ctr., New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
- University of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Background] Burkart GJ, Smaldone GC, Eldon MA, Venkataramanan R, Dauber J, Zeevi A, McCurry K, McKaveney TP, Corcoran TE, Griffith BP, Iacono AT. Lung deposition and pharmacokinetics of cyclosporine after aerosolization in lung transplant patients. Pharm Res. 2003 Feb;20(2):252-6. doi: 10.1023/a:1022275222207. PMID 12636164
- [Background] Iacono AT, Smaldone GC, Keenan RJ, Diot P, Dauber JH, Zeevi A, Burckart GJ, Griffith BP. Dose-related reversal of acute lung rejection by aerosolized cyclosporine. Am J Respir Crit Care Med. 1997 May;155(5):1690-8. doi: 10.1164/ajrccm.155.5.9154878.
- [Background] Keenan RJ, Iacono A, Dauber JH, Zeevi A, Yousem SA, Ohori NP, Burckart GJ, Kawai A, Smaldone GC, Griffith BP. Treatment of refractory acute allograft rejection with aerosolized cyclosporine in lung transplant recipients. J Thorac Cardiovasc Surg. 1997 Feb;113(2):335-40; discussion 340-1. doi: 10.1016/S0022-5223(97)70331-3. PMID 9040628
- [Background] Iacono A, Dauber J, Keenan R, Spichty K, Cai J, Grgurich W, Burckart G, Smaldone G, Pham S, Ohori NP, Yousem S, Williams P, Griffith B, Zeevi A. Interleukin 6 and interferon-gamma gene expression in lung transplant recipients with refractory acute cellular rejection: implications for monitoring and inhibition by treatment with aerosolized cyclosporine. Transplantation. 1997 Jul 27;64(2):263-9. doi: 10.1097/00007890-199707270-00015. PMID 9256185
- [Background] Iacono AT, Johnson BA, Grgurich WF, Youssef JG, Corcoran TE, Seiler DA, Dauber JH, Smaldone GC, Zeevi A, Yousem SA, Fung JJ, Burckart GJ, McCurry KR, Griffith BP. A randomized trial of inhaled cyclosporine in lung-transplant recipients. N Engl J Med. 2006 Jan 12;354(2):141-50. doi: 10.1056/NEJMoa043204. PMID 16407509
- [Background] Iacono AT, Corcoran TE, Griffith BP, Grgurich WF, Smith DA, Zeevi A, Smaldone GC, McCurry KR, Johnson BA, Dauber JH. Aerosol cyclosporin therapy in lung transplant recipients with bronchiolitis obliterans. Eur Respir J. 2004 Mar;23(3):384-90. doi: 10.1183/09031936.04.00058504. PMID 15065826
- [Background] Iacono AT, Keenan RJ, Duncan SR, Smaldone GC, Dauber JH, Paradis IL, Ohori NP, Grgurich WF, Burckart GJ, Zeevi A, Delgado E, O'Riordan TG, Zendarsky MM, Yousem SA, Griffith BP. Aerosolized cyclosporine in lung recipients with refractory chronic rejection. Am J Respir Crit Care Med. 1996 Apr;153(4 Pt 1):1451-5. doi: 10.1164/ajrccm.153.4.8616581.